CLINICAL TRIAL: NCT01141192
Title: The Effect of Vitamin D Supplementation on Glucose Metabolism in Non-Diabetic African American Adults
Acronym: AVIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Jennifer Pederson-White, DO, Medical College of Georgia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0910091
Record Dates: First submitted 2010-06-04; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes
Keywords: vitamin D status; 25-OH D; ionized calcium; fasting glucose; hemoglobin A1c; fasting insulin; glucose metabolism; HOMA index; blood lipids; type 2 diabetes; PTH; adiposity; body fat percentage; dual energy x-ray absorptiometry; pulse wave velocity; arterial stiffness; flow-mediated dilation; African American; inflammatory markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplement (Active Comparator): 60,000 IU vitamin D3 oral supplement provided every four weeks at weeks 0, 4, 8, and 12 in the form of one 50,000 and two 5,000 IU vitamin D3 supplements in gelcap form.
  Interventions: Dietary Supplement: vitamin D3, cholecalciferol
- Sugar Pill (Placebo Comparator): Inactive placebo tablets identical in appearance to the active comparator provided every four weeks at weeks 0,4,8,and 12.
  Interventions: Dietary Supplement: Inactive comparator

INTERVENTIONS:
Dietary Supplement: vitamin D3, cholecalciferol — 1 gelcap of 50,000 IU vitamin D3 plus 2 gelcaps of 5,000 IU vitamin D3 each; a total of 60,000 IU vitamin D3 dosed four weeks apart at weeks 0, 4, 8, and 12 of the 16 week study.
  Arms: Vitamin D3 supplement
Dietary Supplement: Inactive comparator — The inactive comparator dose provided was identical in appearance to the active comparator but contained no vitamin D3
  Arms: Sugar Pill

SUMMARY:
Type 2 diabetes is more common among African Americans than Caucasians. African Americans are also at a higher risk for lower levels of vitamin D compared to other ethnic groups. The investigators don't yet know if there is a connection between not having enough vitamin D and type 2 diabetes in African Americans. Researchers have found that the less vitamin D Caucasians had the higher the chance they would have type 2 diabetes but it is less clear if this is the case for African Americans. The investigators want to better understand how vitamin D status and diabetes risk are linked in African Americans. Also, the investigators want to see if supplementation with vitamin D will improve your blood pressure, blood sugar, & insulin. All of these are in some way related to diabetes. The investigators want to measure changes in blood sugar & blood pressure in people who do not have diabetes with the hope of learning new information to help treat those that do have diabetes.

The investigators hypothesize that vitamin D status is related to diabetes risk measured by hemoglobin A1c (a test of glucose level over time), fasting glucose and insulin in non-diabetic African American adults and that body weight status may affect vitamin D status in response to vitamin D supplements compared to placebo.

DETAILED DESCRIPTION:
Participants will be randomly assigned to receive either a 60,000 IU vitamin D3 supplement every four weeks or an inactive placebo. All investigators and the participants will be blinded to the assignment group of each participant until all testing is completed.

ELIGIBILITY:
Inclusion Criteria:

* African American by self-report
* In good health

Exclusion Criteria:

* Diagnosis of diabetes
* Health problems/medication affecting calcium and/or vitamin D metabolism
* Current use of vitamin/mineral/herbal/nutritional supplements
* Inability to swallow pills
* Pregnancy

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Fasting glucose level before, mid-way through, and after the vitamin D3 supplement or placebo trial. | 16 weeks

SECONDARY OUTCOMES:
Serum 25-OH D levels in response to vitamin D3 supplement or placebo across a range of adiposity | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Dong, MD, PhD, Study Director — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States

REFERENCES:
- [Background] Liu E, Meigs JB, Pittas AG, McKeown NM, Economos CD, Booth SL, Jacques PF. Plasma 25-hydroxyvitamin d is associated with markers of the insulin resistant phenotype in nondiabetic adults. J Nutr. 2009 Feb;139(2):329-34. doi: 10.3945/jn.108.093831. Epub 2008 Dec 23. PMID 19106328
- [Background] Pittas AG, Dawson-Hughes B. Vitamin D and diabetes. J Steroid Biochem Mol Biol. 2010 Jul;121(1-2):425-9. doi: 10.1016/j.jsbmb.2010.03.042. Epub 2010 Mar 18. PMID 20304061
- [Background] Voidonikola PT, Stamatelopoulos KS, Alevizaki M, Kollias GE, Zakopoulos NA, Lekakis JP, Anastasiou E, Theodorakis MJ, Pittas AG, Papamichael CM. The association between glycemia and endothelial function in nondiabetic individuals: the importance of body weight. Obesity (Silver Spring). 2008 Dec;16(12):2658-62. doi: 10.1038/oby.2008.431. Epub 2008 Oct 9. PMID 18846051
- [Background] Liu E, Meigs JB, Pittas AG, Economos CD, McKeown NM, Booth SL, Jacques PF. Predicted 25-hydroxyvitamin D score and incident type 2 diabetes in the Framingham Offspring Study. Am J Clin Nutr. 2010 Jun;91(6):1627-33. doi: 10.3945/ajcn.2009.28441. Epub 2010 Apr 14. PMID 20392893
- [Derived] Zhu H, Guo D, Li K, Pedersen-White J, Stallmann-Jorgensen IS, Huang Y, Parikh S, Liu K, Dong Y. Increased telomerase activity and vitamin D supplementation in overweight African Americans. Int J Obes (Lond). 2012 Jun;36(6):805-9. doi: 10.1038/ijo.2011.197. Epub 2011 Oct 11. PMID 21986705